CLINICAL TRIAL: NCT02892734
Title: A Phase II Window of Opportunity Trial of Ipilimumab and Nivolumab in Metastatic Recurrent HER2- Inflammatory Breast Cancer (IBC) The Win Trial
Brief Title: Ipilimumab and Nivolumab in Treating Patients With Recurrent Stage IV HER2 Negative Inflammatory Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Northwestern University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16B07; STU00203191 (CTRP (Clinical Trial Reporting Program)); NU 16B07 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-01038 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-06

CONDITIONS: HER2/Neu Negative; Recurrent Inflammatory Breast Carcinoma; Stage IV Breast Cancer; Stage IV Inflammatory Breast Carcinoma
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes Q2W and ipilimumab IV over 90 minutes Q6W in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
The purpose of this research study is to look at the efficacy (the effect on tumor) and the safety (the effect on body) of the study drugs when given as a combination in patients with metastatic recurrent epidermal growth factor receptor 2 (HER2) negative inflammatory breast cancer. This is a phase II study of 2 drugs used in combination: nivolumab and ipilimumab. The combination of these drugs is already approved by the Food and Drug Administration (FDA) to treat advanced melanoma (a type of skin cancer). Nivolumab and ipilimumab are not approved by the FDA for patients with metastatic recurrent HER2 negative inflammatory breast cancer, hence the treatment is considered experimental or investigational.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine progression free survival (PFS) in patients with newly recurrent HER2 negative inflammatory breast cancer (IBC) treated with nivolumab and ipilimumab according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.

SECONDARY OBJECTIVES:

I. To assess the overall response rate (ORR) and clinical benefit rate (CBR) according to RECIST criteria v1.1, in patients with recurrent IBC treated with nivolumab and ipilimumab.

II. To assess overall survival in patients with recurrent HER2 negative IBC treated with nivolumab and ipilimumab.

III. To assess the safety and tolerability of nivolumab and ipilimumab in patients with recurrent IBC according to the National Cancer Institute Common Terminology Criteria for Adverse Events v 4.03.

TERTIARY OBJECTIVES:

I. To assess the predictive value of baseline iSCORE and programmed cell death 1 ligand 1 (PDL-1) expression using archival tissue samples as well as any standard of care tissue obtained during study treatment.

II. To assess the predictive value of circulating cell-free tumor DNA (ctDNA) and immune signature by exosome analysis using blood samples at baseline.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes every 2 weeks (Q2W) and ipilimumab IV over 90 minutes every 6 weeks (Q6W) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 weeks for 12 weeks, and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV breast carcinoma with a previous clinical diagnosis of IBC based on the presence of inflammatory changes in the involved breast, such as diffuse erythema and edema (peau d'orange), with or without an underlying palpable mass involving the majority of the skin of the breast; pathological evidence of dermal lymphatic invasion should be noted but is not required for diagnosis
* Patients must have local or metastatic recurrence of IBC after prior surgery
* Patients must have a metastatic tumor negative for HER2; the lack of HER2 overexpression by immunohistochemistry (IHC), is defined as 0 or 1+ where as hyperexpression is defined as 3+; if equivocal IHC, 2+, the tumor must be non-gene amplified by fluorescence in situ hybridization (FISH) performed upon the primary tumor or metastatic lesion (ratio < 2 and HER2 copy number < 4)
* Patients may have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1 OR non-measurable tumors; NOTE: Non-measurable tumors are small lesions (longest diameter < 10mm or pathological lymph nodes with >= 10 to < 15 mm short axis); bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonitis, inflammatory breast disease, and abdominal masses (not followed by computed tomography [CT] or magnetic resonance imaging [MRI]) are considered as non-measurable
* Patients must be in consideration for 1st line systemic therapy for recurrent IBC; NOTE: Patients must not have received chemotherapy in the metastatic setting, but adjuvant treatment after surgery is acceptable
* Patients must have confirmed availability of archival or freshly biopsied tumor tissue meeting protocol-defined specifications prior to study enrollment
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) status of 0-1; ECOG performance status 2 and 3 will be allowed only if decline in performance status is thought to be directly secondary to breast cancer disease burden by treating physician
* Patients must have adequate organ and bone marrow function within 14 days prior to registration, as defined below:
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL, regardless of transfusion or growth factor support
* Platelets >= 100,000/mcl, regardless of transfusion or growth factor support
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert syndrome or liver metastasis who can have total bilirubin < 3.0 x ULN)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/ alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 x upper limit of normal (ULN) (or =< 5 times ULN in case of liver metastasis)
* Serum creatinine of < 3.0 x ULN (upper limit of normal)
* Patients with history of central nervous system (CNS) metastases are eligible if CNS disease has been stable for at least 6 weeks prior to study registration in the opinion of the investigator and do not require corticosteroids (of any dose) for symptomatic management; NOTE: Patients are not required to have CNS imaging prior to study entry
* Females of childbearing potential (FOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours of registration

NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

  * FOCBP and men who are sexually active with FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment and the designated post-treatment period
  * Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients must not have had chemotherapy or radiotherapy within 4 weeks prior to study registration
* Patients who already received chemotherapy for recurrent metastatic IBC are not eligible
* Patients who have not recovered to =< grade 1 from adverse events due to agents administered more than 4 weeks earlier are not eligible
* Patients may not be receiving any other investigational agents
* Patients who have had prior exposure to immune checkpoint inhibitors are not eligible; please contact principal investigator, Ricardo Costaat 312-472-1234 for specific questions on potential interactions

  * Programmed cell death protein 1 (PD-1) monoclonal antibody: pembrolizumab, pidilizumab, MEDI-0680, anti-PD-1 fusion protein AMP-224 (AMP-224), anti-PD-1 checkpoint inhibitor PF-06801591 (PF-06801591), anti-PD-1 monoclonal antibody BGB-A317 (BGB-A317), anti-PD-1 monoclonal antibody PDR001 (PDR001), anti-PD-1 monoclonal antibody REGN2810 (REGN2810), anti-PD-1 monoclonal antibody SHR-1210 (SHR-1210)
  * PD-L1 monoclonal antibody: durvalumab, avelumab, anti-PD-L1 monoclonal antibody MDX-1105 (MDX-1105), atezolizumab, zirconium Zr 89-labeled anti-PD-L1 monoclonal antibody MPDL3280A (MPDL3280A)
  * Cytotoxic T-lymphocyte protein 4 (CTLA4) monoclonal antibody: tremelimumab, abatacept
  * Tumor necrosis factor receptor superfamily member 4 (OX40): agonistic anti-OX40 monoclonal antibody MEDI6383 (MEDI6383), agonistic anti-OX40 monoclonal antibody MEDI6469 (MEDI6469), anti-OX40 monoclonal antibody MEDI0562 (MEDI0562), oxelumab, anti-OX40 antibody PF-04518600 (PF-04518600)
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded; these include but are not limited to patients with a history of:

  * Immune related neurologic disease
  * Multiple sclerosis
  * Autoimmune (demyelinating) neuropathy
  * Guillain-Barre syndrome
  * Myasthenia gravis
  * Systemic autoimmune disease such as systemic lupus erythematosus (SLE)
  * Connective tissue diseases
  * Scleroderma
  * Inflammatory bowel disease (IBD)
  * Crohn's
  * Ulcerative colitis
  * Patients with a history of toxic epidermal necrolysis (TEN)
  * Stevens-Johnson syndrome
  * Anti-phospholipid syndrome
  * NOTE: Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Ongoing or active infection (including minor localized infections) requiring oral or IV treatment
  * Symptomatic congestive heart failure, defined as a clinical syndrome resulting from any structural or functional cardiac disorder that impairs the ability of the ventricle to fill with or eject blood
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients should not have any condition requiring systemic treatment with corticosteroids (< 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug; NOTE: Inhaled or topical steroids and adrenal replacement steroid doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; a brief (less than 3 weeks) course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by a contact allergen) is permitted
* Female patients who are pregnant or nursing are not eligible
* No other prior malignancy is allowed except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Or any other cancer from which the patient has been disease free for at least three years
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) is not permitted
* Any known positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection is not permitted
* Patients who have received a live attenuated vaccine within 30 days are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Costa, M.D., M.Sc., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on September 5, 2017 with a total accrual goal of 29. The first patient started treatment October 18, 2017. The study was closed permanently January 21 2019 with 3 patients treated on study.
Groups:
- Treatment (Nivolumab, Ipilimumab): Patients receive nivolumab 240mg IV over 30 minutes Q2W for the first 16 weeks then 480mg IV every 4 weeks thereafter. Patients will Ipilimumab 1mg/kg IV over 90 minutes Q6W in the absence of disease progression or unacceptable toxicity. 1 Cycle = 12 weeks. Scans every 12 weeks for disease assessment.
  Ipilimumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
Period: Treatment on Study
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Started | 3
Completed 1st Cycle/Response at 12 Weeks | 1
Went on to Start Cycle 2 | 1
Completed | 1
Not Completed | 2
Not completed — Progressive Disease | 2
Period: Follow up for 2 Years
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Started (All patients that are treated with at least one dose of study drug go into follow-up.) | 3
Completed | 0
Not Completed | 3
Not completed — Death | 2
Not completed — Study closed early | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS in patients with newly recurrent HER2 negative IBC treated with nivolumab and ipilimumab as evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 assessed from the date of first study treatment to the date of disease progression or death from any cause, assessed up to 2 years.
Time Frame: Up to 2 years
Population: Data not collected and analyzed as study closed to accrual early due to slow accrual.
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Evaluate the ORR according to RECIST criteria v1.1 in patients with recurrent Inflammatory Breast Cancer (IBC) treated with nivolumab and ipilimumab. ORR will be the number of patients with complete response plus the number of patients with partial response. Patients will have imaging scans every 12 weeks assessed up to 2 years.
  In general:
  Complete Response (CR): Disappearance of all target and non target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 12 weeks from treatment initiation for up to 2 years. Range of cycles patients completed 1-3 cycles (1 cycle =12 weeks)
Population: Sample size was too small for statistical analysis. Data collected shown but should be viewed as incomplete as based off of 1 patient. Only those patients who have measurable disease present at baseline, have received at least one dose of therapy, and have had their disease re-evaluated will be considered evaluable for response.
Measure: Number; unit: patients
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 1
patients | 0

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Evaluate the CBR according to RECIST criteria v1.1 in patients with recurrent Inflammatory Breast Cancer (IBC) treated with nivolumab and ipilimumab. CBR will be the number of patients with complete response plus the number of patients with partial response plus those with stable disease. Patients will have imaging scans every 12 weeks assessed up to 2 years.
  In general:
  Complete Response (CR): Disappearance of all target and non target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: number of patients
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 1
number of patients | 1

4. Secondary Outcome: Overall Survival (OS)
Description: To assess overall survival in patients with recurrent HER2 negative IBC treated with nivolumab and ipilimumab, patients will be followed from the start of treatment until 2 years post-treatment or death, whichever occurs first, and average survival time will be measured.
Time Frame: Up to 2 years
Population: OS was not calculated. Sample size was too small to warrant analysis due to the study closes before accrual was reached. Reported below is the number of patients alive at the time of reporting data (4/12/2019).
Measure: Number; unit: patients
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 3
patients | 1

5. Secondary Outcome: Number of Adverse Events of Nivolumab and Ipilimumab Combination Treatment
Description: Assess the safety and tolerability of nivolumab and ipilimumab in patients with recurrent Inflammatory Breast Cancer (IBC) by measuring the number, frequency, and severity of adverse events according to the National Cancer Institute Common Terminology Criteria Adverse events (CTCAE) v 4.03. AEs that were determined to be at least possibly related to study drug and grade 3-5 are reported.
  In general grading is as follows:
  Grade 1 - mild Grade 2 - moderate Grade 3 - severe Grade 4 - life threatening Grade 5 - fatal
Time Frame: From the initiation of treatment until 12 weeks after study discontinuation. Range of cycles completed by patients 1-3 (1 cycle =12weeks)
Population: Data that was collected is reported.
Measure: Number; unit: Adverse Events
Arm/Group | Treatment (Nivolumab, Ipilimumab)
Number analyzed (Participants) | 3
Adverse Events | 1

6. Other Pre Specified Outcome: iScore
Description: Assess the predictive value of baseline iSCORE using tissue samples.
Time Frame: At baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: PD-L1 Expression Measured in Tissue Samples
Time Frame: At baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: ctDNA Assessed by Exosome Analysis in Blood Samples
Time Frame: At baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Immune Signature Assessed by Exosome Analysis in Blood Samples
Time Frame: At baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from treatment initiation through 12 weeks post last dose of study drug with the range of cycles completed by patients 1 - 3. (1 Cycle = 12 Weeks)
Arm/Group | Treatment (Nivolumab, Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Ipilimumab) (N=3)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient also with Pleural effusion during the event.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient also with left pleural effusion at the time of the event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nivolumab, Ipilimumab) (N=3)
Constipation (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Lymphocyte Count Decreased (Investigations) | 2
Aspartate Aminotransferase Increased (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Study closed due to slow accrual after only 3 patients were treated on study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT02892734/Prot_SAP_000.pdf